CLINICAL TRIAL: NCT06089044
Title: Evaluation of the Efficacy and Safety of Suppressive Therapy With DALBAVANCINE in Device Infections
Acronym: DALBASAT
Status: Completed | Type: Observational
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHT/URC/2023/12
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Prosthesis-related Infections
MeSH Terms: conditions — Prosthesis-Related Infections | interventions — dalbavancin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dalbavancin Injection — Dalbavancin as long-term suppressive therapy.

SUMMARY:
The aim of this retrospective observational study is to evaluate the efficacy of antibiotic therapy with dalbavancin in patients presenting with infection on prosthetic devices. The main questions the study aims to answer are:

What is the proportion of patients with early discontinuation of dalbavancin therapy? What are the reasons for early discontinuation of antibiotic treatment? What adverse events do patients report? The study is based on data collected as part of routine care practices.

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion Criteria:

* Patients with inextricable and/or inoperable osteoarticular or vascular prosthetic material.
* Patients requiring suppressive antibiotic therapy (>6 months) with dalbavancin.

Exclusion Criteria:

* Patients who are protected adult;
* Patients who are minors;
* Patients having expressed their opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for a prosthetic device infection requiring suppressive antibiotic therapy for more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
efficacy of suppressive Dalbavancin therapy | two-year follow-up after initiation of suppressive therapy with Dalbavancin
  Proportion of patients successfully treated with Dalbavancin. The efficacy of suppressive therapy will be defined over a two-year period after initiation of treatment as the combination of the following criteria:
  Clinical control of infection :
  * Absence of local inflammatory signs (erythema, discharge, edema, pain) ;
  * Absence of general signs (hyperthermia: T°>38 or hypothermia T°< 36°);
  Biological control:
  o CRP negative (<5mg/l) ;

CONTACTS AND LOCATIONS:
Locations (1):
- CH Tourcoing, Tourcoing, France

IPD SHARING:
Plan to Share IPD: No